CLINICAL TRIAL: NCT06324513
Title: Adaptation of the Mediterranean Diet Pattern to the Exclusion Diet for Crohn's Disease: Assessment of Efficacy and Tolerability in Pediatric and Adult Patients. Non-profit, Multicenter, Randomized, Controlled Study.
Brief Title: Evaluation of the Efficacy and Tolerability of the Mediterranean Diet Pattern in the Exclusion Diet for Patients With Crohn's Disease.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Paolo Lionetti, Principal Investigator, Meyer Children's Hospital IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Med-CDED
Record Dates: First submitted 2024-02-22; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Med-CDED (Experimental): The Mediterranean Crohn's Disease Exclusion Diet (Med-CDED) is the exclusion diet (CDED) adapted to the Mediterranean diet pattern. The Med-CDED consists of 2 phases in dietary therapy and a maintenance phase: the first phase lasting 8 weeks, the second phase lasting 16 weeks, and the maintenance phase, which for the purposes of the study will last 28 weeks.
  Interventions: Dietary Supplement: Mediterranean Crohn's Disease Exclusion Diet (Med-CDED)
- CDED (Active Comparator): The original Crohn's disease exclusion diet, used as a comparator, is widely employed among first-line treatments in clinical practice for inducing remission in pediatric patients with Crohn's disease
  Interventions: Dietary Supplement: Crohn's disease exclusion diet (CDED)

INTERVENTIONS:
Dietary Supplement: Mediterranean Crohn's Disease Exclusion Diet (Med-CDED) — The Mediterranean Crohn's Disease Exclusion Diet (Med-CDED) is the exclusion diet (CDED) adapted to the Mediterranean diet pattern. The Med-CDED consists of 2 phases in dietary therapy and a maintenance phase: the first phase lasting 8 weeks, the second phase lasting 16 weeks, and the maintenance phase, which for the purposes of the study will last 28 weeks.
  Arms: Med-CDED
Dietary Supplement: Crohn's disease exclusion diet (CDED) — The original Crohn's disease exclusion diet, used as a comparator, is widely employed among first-line treatments in clinical practice for inducing remission in pediatric patients with Crohn's disease.
  Arms: CDED

SUMMARY:
The proposed study aims to assess the efficacy and tolerability of adapting the CDED to the Mediterranean diet pattern, without compromising its key principles, namely the exclusion of ultra-processed foods with potential pro-inflammatory effects on the intestines. The decision to modify the CDED according to the characteristics of the Mediterranean diet pattern and to evaluate the potential of this modified version of the exclusion diet for Crohn's disease in terms of efficacy and tolerability are the main objectives of this study.

These objectives are driven not only by scientific evidence regarding the anti-inflammatory potential and protective role against chronic-degenerative diseases demonstrated by the Mediterranean diet but also to allow for greater adherence to Italian dietary traditions and improve compliance with the dietary regimen.

Furthermore, to date, there are no comprehensive multi-omic investigations integrating dietary data with microbiome, metabolome, and transcriptome profiles that can demonstrate the effect of the CDED at "omic" levels. A very recent study on pediatric patients shows interesting results regarding differential profiles of fecal metabolites after administration of CDE or NEE in different weeks of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a stable diagnosis of Crohn's disease according to the criteria of the ECCO/ESPGHAN guidelines.
* Patients with a new diagnosis of the disease or with a disease diagnosed no more than three years ago, receiving stable pharmacological therapy for at least 2 months with immunomodulators (thiopurines, methotrexate, azathioprine) or biologic drugs who have experienced a disease relapse and require reinduction of remission.
* Mild to moderate disease activity assessed by the wPCDAI score between 12.5-57.5 in the pediatric population and a Harvey-Bradshaw Index ranging from 5 to 16 for the adult population.
* Biochemical evidence of active intestinal inflammation at enrollment, assessed by inflammatory markers such as C-reactive protein (CRP) levels ≥ 0.5 mg/dl or fecal calprotectin ≥ 150 mg/g.
* Ability to provide biological samples (stool and blood samples).

Exclusion Criteria:

* Monogenic disease;
* Disease with fibrostenotic or penetrating phenotype;
* Complex perianal fistulizing disease not completely in remission;
* Patients with ileostomy or who have undergone intestinal resection or colectomy;
* Patients currently undergoing other nutritional therapy (e.g., exclusive enteral nutrition) or who have undergone it in the last month;
* Patients not on stable therapy with immunomodulators or biologic drugs or who started therapy with thiopurines less than 4 weeks before enrollment, or methotrexate less than 8 weeks before enrollment;
* Patients with recent use of systemic steroids in the four weeks before enrollment or recent initiation or dose adjustment phase of therapy with immunomodulators (e.g., azathioprine, 6-mercaptopurine, or methotrexate) or biologic drugs;
* Pregnancy;
* Vegan or vegetarian patients;
* Celiac disease.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-07-27 (Estimated); Study Completion 2025-10-27 (Estimated)

PRIMARY OUTCOMES:
Clinical response to the first phase of diet | 8 weeks
  reduction of 12.5 points in the wPCDAI score.
Clinical remission rate | 8 weeks
  wPCDAI score must be <12.5 points after the first phase of diet
Adherence rate to the Med-CDED diet and comparison to the original CDED both in pediatric and adult cohort | Anytime during the study
  Adherence rate will be assessed by adherence questionnaire score or by considering the number of patients who refuse the diet
Clinical remission rate in adult patients at the end of phase I of diet | 8 weeks
  Clinical remission will be assessed by HBI < 5 points

SECONDARY OUTCOMES:
Transmural response of the thickness of the intestinal loops both in pediatric and adult cohort | 0, 8, 24, 38 and 52 weeks
  The thickness of intestinal loops will be assess by using ultrasound
Assessment of the reduction or normalization of inflammation markers both in pediatric and adult cohort | 8 weeks
  ESR, CPR and fecal calprotectin will be measured at the end of phase I of the diet
Assessment of clinical remission rate at the end of Phase II of the Med-CDED diet and comparision with the original CDED both in pediatric and adult cohort | 24 weeks
  Assessment of clinical remission rate at Phase II of both diet protocols
Assessment of clinical remission rate at the end of Phase III of the Med-CDED diet and comparision with the original CDED both in pediatric and adult cohort | 52 weeks
  Assessment of clinical remission rate at Phase III of both diet protocols
Endoscopic response rate obtained at 6 months both in pediatric and adult cohort | 0 and 26 weeks
  The assessment will be performed in a subgroup of partecipants that will recive endoscopy at baseline and after 6 months
Assessment of the modification of the intestinal microbiota composition (trough alpha and beta diversity) at the end of the various phases of the Med-CDED and comparison with the original CDED both in pediatric and adult cohort | 52 weeks
  Bioinformatic analysis of the composition of the intestinal microbiota will be performed after extraction of bacterial genomic DNA from the collected faecal samples and NGS sequencing with the Illumina MiSeq platform. These analyses will allow taxonomic identification of theintestinal microbial communities in each patient. Indices of microbial richness and biodiversity (Chao index, Shannon and Simpson index) will be calculated, and principal coordinate (PCoA) and multidimensional (NMDS) analyses will be performed to assess variability in microbial composition between the various phases of the dietary intervention.
Assessment of the metabolome profiles at the end of the various phases of the Med-CDED and comparison with the original CDED both in pediatric and adult cohort | 52 weeks
  faecal metabolome will be carried out by gas chromatography and mass spectrometry analysis. The identification of differentially abundant metabolites will be carried out by comparing profiles at various stages of the dietary intervention.
Assessment of the trascriptome profiles at the end of the various phases of the Med-CDED and comparison with the original CDED both in pediatric and adult cohort | 52 weeks
  Transcriptome investigation of blood samples, gene expression profiles of the individual's RNA, will be identified by NGS sequencing techniques. Transcriptomic analysis will be performed in R using the DESeq2 package
Ability to maintain a healthy and balanced diet and patient satisfaction with the treatment both in pediatric and adult cohortreceived | Anytime during the study
  Ability to maintain a healthy and balanced diet and patient satisfaction with the treatment recived assessed with nutritional questionnair

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Meyer Children's Hospital IRCCS, Florence
  - Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - Università La Sapienza di Roma, Roma

IPD SHARING:
Plan to Share IPD: No